CLINICAL TRIAL: NCT06253663
Title: A Phase 2 Multicenter Study Evaluating the Safety and the Efficacy of KTE-X19 in Adult Japanese Subjects With Relapsed/Refractory Mantle Cell Lymphoma or Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia
Brief Title: Study of KTE-X19 in Adult Japanese Participants With Relapsed/Refractory Mantle Cell Lymphoma or Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia
Acronym: JKART-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-472-0149
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Mantle Cell Lymphoma; Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — brexucabtagene autoleucel; Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: Participant will be enrolled into the appropriate cohort depending on the type of disease in the two cohorts: r/r Mantle Cell Lymphoma (MCL) or r/r B-precursor Acute Lymphoblastic Leukemia(B-ALL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MCL Cohort- KTE-X19 (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV lymphodepletion chemotherapy for 3 days followed by KTE-X19 administered intravenously at a target dose of 2 x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) T cells/kg on Day 0.
  For participants weighing ≥ 100 kg, a maximum flat dose of 2 x 10^8 anti-CD19 CAR T cells will be administered.
  Interventions: Drug: KTE-X19; Drug: Cyclophosphamide; Drug: Fludarabine
- ALL Cohort- KTE-X19 (Experimental): Participants will receive cyclophosphamide 900 mg/m^2/day intravenously (IV) for 1 day and fludarabine 25 mg/m^2/day IV lymphodepletion chemotherapy for 3 days followed by KTE-X19 administered intravenously at a target dose of 1 x 10^6 19 CAR T cells/kg on Day 0.
  For participants weighing ≥ 100 kg, a maximum flat dose of 1 x 10^8 anti-CD19 CAR T cells will be administered.
  Interventions: Drug: KTE-X19; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: KTE-X19 — A single infusion of chimeric antigen receptor (CAR) T cells
  Other Names: Tecartus
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously

SUMMARY:
The goal of this clinical study is to learn more about KTE-X19, and how safe and effective it is in adult Japanese participants with relapsed/refractory (r/r) Mantle Cell Lymphoma (MCL) or r/r B-precursor Acute Lymphoblastic Leukemia (B-ALL).

The primary objectives of this study are to evaluate the efficacy of KTE-X19, as measured by:

* Objective response rate (ORR) per investigator assessment, in adult Japanese participants with r/r MCL
* Overall complete remission (OCR) defined as complete remission (CR) and complete remission with incomplete hematologic recovery (CRi) per investigator assessment, in adult Japanese participants with r/r ALL

DETAILED DESCRIPTION:
After completing at least 24 months in the study, all participants who received an infusion of KTE-X19 will be transitioned to a separate long-term follow-up (LTFU) study (KT-US-982-5968) to complete the remainder of the 15-year follow-up assessments.

ELIGIBILITY:
Key Inclusion Criteria:

MCL Cohort:

* Pathologically confirmed MCL, with documentation of either overexpression of cyclin D1 or presence of t(11;14)
* Up to 5 prior regimens for MCL. Prior therapy must have included:

  * Anthracycline-, bendamustine-, or high-dose cytarabine- containing chemotherapy, and
  * Anti-CD20 monoclonal antibody therapy, and
  * Bruton's tyrosine kinase inhibitor (BTKi)
* Relapsed or refractory disease, defined by the following:

  * Disease progression after last regimen, or
  * Refractory disease is defined failure to achieve partial response (PR) or complete remission (CR) to the last regimen
* At least 1 measurable lesion. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy

  * If the only measurable disease is lymph node disease, at least 1 lymph node should be ≥ 2 cm

ALL Cohort:

* Relapsed or refractory B-ALL defined as one of the following:

  * Relapsed or refractory disease after one line of systemic therapy;

    * Primary refractory, or
    * First relapse if first remission ≤ 12 months
  * Relapsed or refractory disease after two or more lines of systemic therapy
  * Relapsed or refractory disease after allogeneic transplant provided individuals is at least 100 days from SCT at the time of enrollment and off of immunosuppressive medications for at least 4 weeks prior to enrollment
* Morphological disease in the bone marrow (> 5% blasts)
* Individuals with Philadelphia-positive (Ph+) disease are eligible if they are intolerant to tyrosine kinase inhibitor (TKI) therapy, or if they have relapsed/refractory disease despite treatment with at least 2 different TKIs

Key Exclusion Criteria:

MCL Cohort:

* History of malignancy other than nonmelanomatous skin cancer or carcinoma in situ (eg, cervix, bladder, breast) unless disease-free for at least 3 years
* Autologous SCT (autoSCT) within 6 weeks of planned KTE-X19 infusion
* History of alloSCT with the exception of individuals with no donor cells detected on chimerism > 100 days after alloSCT
* Prior CD19 targeted therapy
* Prior CAR therapy or other genetically modified T-cell therapy
* History of hypersensitivity to any of the ingredients of KTE-X19 or to any of the animal-derived ingredients (bovine and rodent) used in the manufacturing process of KTE-X19

ALL Cohort:

* Diagnosis of Burkitt's leukemia/lymphoma according to World Health Organization (WHO) classification or chronic myelogenous leukemia lymphoid blast crisis
* History of malignancy other than non-melanoma skin cancer or carcinoma in situ (eg, cervix, bladder, breast) unless disease free for at least 3 years
* History of hypersensitivity to any of the ingredients of KTE-X19 or to any of the animal-derived ingredients (bovine and rodent) used in the manufacturing process of KTE-X19

Note: Other protocols defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
MCL Cohort: Objective Response Rate (ORR) Per Investigator Assessment | Up to 24 months
  ORR is defined as the incidence of a complete remission (CR) or a partial remission (PR) per the Lugano Classification.
ALL Cohort: Overall Complete Remission (OCR) Rate | Up to 24 months
  OCR rate is defined as the percentage of participants achieving CR/complete remission with incomplete hematologic recovery (CRi) per investigator assessment.

SECONDARY OUTCOMES:
MCL Cohort: Duration of Response (DOR) | Up to 24 months
  DOR is defined as time from first objective response to disease progression per indication specific response criteria or death from any cause.
MCL Cohort: Best Objective Response (BOR) | Up to 24 months
  BOR is defined as the incidence of CR, PR, Stable disease (SD) or progressive disease (PD) or unevaluable as best response to treatment.
MCL Cohort: Progression-Free Survival (PFS) | Up to 24 months
  PFS is defined as time from enrollment or KTE-X19 infusion to disease progression per indication specific response criteria or death from any cause.
MCL Cohort: Levels of Cytokines in Serum | Up to Day 28
ALL Cohort: Minimal Residual Disease (MRD) Negativity Rate | Up to 24 months
  The incidence of a minimal residual disease response (MRD-). MRD- is defined as MRD < 10^-6 per the standard assessment.
ALL Cohort: Allogeneic Stem Cell Transplant (alloSCT) rate | Up to 24 months
  The percentage of participants receiving alloSCT as the 1st next therapy after KTE-X19 infusion.
ALL Cohort: Relapse-Free Survival (RFS) | Up to 24 months
  RFS is defined as the time from enrollment or KTE-X19 infusion date to the date of disease relapse or death from any cause.
ALL Cohorts: DOR | Up to 24 months
  DOR is defined as the time between their first complete remission (CR or CRi) to relapse or any death in the absence of documented relapse.
MCL and ALL Cohort: Levels of Anti-Cluster of Differentiation 19 (Anti-CD19) CAR T Cells in Blood | Up to 24 months
MCL and ALL Cohorts: Percentages of Participants Experiencing Treatment-emergent Adverse Event (TEAEs), Serious Adverse Event (SAEs) and Deaths | First infusion date up to 24 months
MCL and ALL Cohorts: Overall Survival (OS) | Up to 24 months
  OS is defined as the time from enrollment or KTE-X19 infusion to death from any cause.
MCL and ALL Cohorts: Percentage of Participants Experiencing Clinically Significant Changes in Safety Laboratory Values | First infusion date up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (9):
- Japan (9):
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Kyoto University Hospital, Kyoto
  - Tohoku University Hospital, Miyagi
  - Okayama University Hospital, Okayama
  - National Cancer Center Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06253663